CLINICAL TRIAL: NCT05382754
Title: Home Sleep Apnea Testing Compared to In-lab Polysomnography for the Evaluation of Obstructive Sleep Apnea in Children
Brief Title: Home Apnea Testing in CHildren Trial
Acronym: HATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 21-019533; 1R61HL162839-01 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Sleep Apnea, Obstructive; Sleep Disorder; Sleep Apnea Syndromes; Sleep Disturbance
Keywords: obstructive sleep apnea; home sleep apnea testing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders; Sleep Apnea Syndromes; Parasomnias

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the initial test (home sleep apnea test or polysomnography) and then complete the alternate test within one week.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators will be masked as to the order of the two sleep tests
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- HSAT first (Experimental): Participants will be randomized to undergo HSAT before receiving their clinical, in-lab polysomnography
  Interventions: Diagnostic Test: Home sleep apnea test
- PSG first (Active Comparator): Participants will be randomized to undergo HSAT after receiving their clinical, in-lab polysomnography.
  Interventions: Diagnostic Test: In-lab polysomnography

INTERVENTIONS:
Diagnostic Test: Home sleep apnea test — Level II home sleep apnea testing evaluates for obstructive sleep apnea in the home environment with parental supervision.
  Other Names: NOX A1; HSAT
  Arms: HSAT first
Diagnostic Test: In-lab polysomnography — Overnight sleep study in the sleep laboratory with continuous monitoring by clinical staff.
  Other Names: PSG
  Arms: PSG first

SUMMARY:
This clinical trial will compare home sleep apnea testing with the gold standard in-lab polysomnography in terms of 1) accuracy, 2) therapeutic decision-making, and 3) parent/child acceptability in children referred for evaluation of obstructive sleep apnea.

DETAILED DESCRIPTION:
In-lab attended polysomnography (PSG) is recommended for the diagnosis of obstructive sleep apnea (OSA) in children, but testing is limited by high cost and limited facilities. 90% of children who undergo adenotonsillectomy to treat OSA never have the diagnosis made by PSG. Home sleep apnea testing (HSAT) is an accepted means of evaluating adults for OSA. However, in children there is insufficient evidence comparing HSAT to PSG, so it is not currently recommended in the pediatric population. This single-center comparative effectiveness trial will compare the diagnostic accuracy of HSAT with PSG and will assess the agreement in therapeutic decision-making between the two tests and parent- and child-reported acceptability of HSAT and preference of test.

Participants will be randomized to the initial test (HSAT or PSG) and then complete the alternate test within one week. Off-site investigators who are pediatric sleep medicine physicians will provide a therapeutic decision based on clinical data and either HSAT or PSG data, and families will complete questionnaires assessing acceptability of HSAT and preference between the two tests.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children age 5-12 years old inclusive
* Referred for diagnostic PSG at the Children's Hospital of Philadelphia (CHOP) Sleep Laboratory for evaluation of OSA as part of clinical care
* Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

* Children without Down syndrome who have had a PSG within 3 years of enrollment
* Children with Down syndrome who have had a PSG within 1 year of enrollment.
* Children with a history of hypoventilation or hypoxemia or who require supplemental oxygen or positive airway pressure during sleep
* Children with a tracheostomy or tracheocutaneous fistula
* Children who live in a facility without their parent

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 317 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with diagnosis of OSA on both HSAT and PSG | 2 weeks
  Obstructive sleep apnea (OSA) defined as an obstructive apnea hypopnea index of greater than 2 events/hour on both home sleep apnea test (HSAT) and polysomnography (PSG).

SECONDARY OUTCOMES:
Association between therapeutic decision from HSAT compared to PSG | 2 weeks
  Logistic regression will compare therapeutic decision (conservative management versus active treatment) from home sleep apnea test (HSAT) or polysomnography (PSG) by investigator blinded to the result of the alternate test.
Proportion of participants who prefer HSAT to PSG | 2 weeks
  Parents of participants will report which test they prefer and both parent and child will report acceptability of home sleep apnea test
Correlation between obstructive apnea hypopnea index (OAHI) of HSAT compared to PSG | 2 weeks
  Obstructive apnea hypopnea index will be assessed as a continuous variable with polysomnography (PSG) assigned as the reference test compared to home sleep apnea test (HSAT).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Cielo, DO, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) will be made available upon reasonable request after completion of the trial and publication of the primary results. Access will be provided following review and approval of a research proposal, with a signed data use agreement and any necessary ethical approvals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It is anticipated that the data from this study will be used to guide future evidence-based guidelines regarding the evaluation of OSA in children. We will submit to the National Library of Medicine's PubMed Central an electronic version of the final, peer-reviewed manuscripts upon acceptance for publication, to be made publicly available no later than 12 months after the official date of publication.

REFERENCES:
- [Background] Marcus CL, Traylor J, Biggs SN, Roberts RS, Nixon GM, Narang I, Bhattacharjee R, Davey MJ, Horne RS, Cheshire M, Gibbons KJ, Dix J, Asztalos E, Doyle LW, Opie GF, D'ilario J, Costantini L, Bradford R, Schmidt B. Feasibility of comprehensive, unattended ambulatory polysomnography in school-aged children. J Clin Sleep Med. 2014 Aug 15;10(8):913-8. doi: 10.5664/jcsm.3970. PMID 25126039
- [Background] Goodwin JL, Enright PL, Kaemingk KL, Rosen GM, Morgan WJ, Fregosi RF, Quan SF. Feasibility of using unattended polysomnography in children for research--report of the Tucson Children's Assessment of Sleep Apnea study (TuCASA). Sleep. 2001 Dec 15;24(8):937-44. doi: 10.1093/sleep/24.8.937. PMID 11766164
- [Background] Guilleminault C, Lee JH, Chan A. Pediatric obstructive sleep apnea syndrome. Arch Pediatr Adolesc Med. 2005 Aug;159(8):775-85. doi: 10.1001/archpedi.159.8.775. PMID 16061787
- [Background] Bixler EO, Vgontzas AN, Lin HM, Liao D, Calhoun S, Vela-Bueno A, Fedok F, Vlasic V, Graff G. Sleep disordered breathing in children in a general population sample: prevalence and risk factors. Sleep. 2009 Jun;32(6):731-6. doi: 10.1093/sleep/32.6.731. PMID 19544748
- [Background] Li AM, So HK, Au CT, Ho C, Lau J, Ng SK, Abdullah VJ, Fok TF, Wing YK. Epidemiology of obstructive sleep apnoea syndrome in Chinese children: a two-phase community study. Thorax. 2010 Nov;65(11):991-7. doi: 10.1136/thx.2010.134858. PMID 20965935
- [Background] Horne RS, Yang JS, Walter LM, Richardson HL, O'Driscoll DM, Foster AM, Wong S, Ng ML, Bashir F, Patterson R, Nixon GM, Jolley D, Walker AM, Anderson V, Trinder J, Davey MJ. Elevated blood pressure during sleep and wake in children with sleep-disordered breathing. Pediatrics. 2011 Jul;128(1):e85-92. doi: 10.1542/peds.2010-3431. Epub 2011 Jun 27. PMID 21708802
- [Background] Marcus CL, Moore RH, Rosen CL, Giordani B, Garetz SL, Taylor HG, Mitchell RB, Amin R, Katz ES, Arens R, Paruthi S, Muzumdar H, Gozal D, Thomas NH, Ware J, Beebe D, Snyder K, Elden L, Sprecher RC, Willging P, Jones D, Bent JP, Hoban T, Chervin RD, Ellenberg SS, Redline S; Childhood Adenotonsillectomy Trial (CHAT). A randomized trial of adenotonsillectomy for childhood sleep apnea. N Engl J Med. 2013 Jun 20;368(25):2366-76. doi: 10.1056/NEJMoa1215881. Epub 2013 May 21. PMID 23692173
- [Background] Gozal D, Crabtree VM, Sans Capdevila O, Witcher LA, Kheirandish-Gozal L. C-reactive protein, obstructive sleep apnea, and cognitive dysfunction in school-aged children. Am J Respir Crit Care Med. 2007 Jul 15;176(2):188-93. doi: 10.1164/rccm.200610-1519OC. Epub 2007 Mar 30. PMID 17400731
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Das S, Mindell J, Millet GC, Ofer D, Beck SE, Mason TB, Brooks LJ, Traylor J, Marcus CL. Pediatric polysomnography: the patient and family perspective. J Clin Sleep Med. 2011 Feb 15;7(1):81-7. PMID 21344042
- [Background] Rosen IM, Kirsch DB, Chervin RD, Carden KA, Ramar K, Aurora RN, Kristo DA, Malhotra RK, Martin JL, Olson EJ, Rosen CL, Rowley JA; American Academy of Sleep Medicine Board of Directors. Clinical Use of a Home Sleep Apnea Test: An American Academy of Sleep Medicine Position Statement. J Clin Sleep Med. 2017 Oct 15;13(10):1205-1207. doi: 10.5664/jcsm.6774. PMID 28942762
- [Background] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- [Background] Kuna ST, Gurubhagavatula I, Maislin G, Hin S, Hartwig KC, McCloskey S, Hachadoorian R, Hurley S, Gupta R, Staley B, Atwood CW. Noninferiority of functional outcome in ambulatory management of obstructive sleep apnea. Am J Respir Crit Care Med. 2011 May 1;183(9):1238-44. doi: 10.1164/rccm.201011-1770OC. Epub 2011 Jan 21. PMID 21471093
- [Background] Berry RB, Hill G, Thompson L, McLaurin V. Portable monitoring and autotitration versus polysomnography for the diagnosis and treatment of sleep apnea. Sleep. 2008 Oct;31(10):1423-31. PMID 18853940
- [Background] Skomro RP, Gjevre J, Reid J, McNab B, Ghosh S, Stiles M, Jokic R, Ward H, Cotton D. Outcomes of home-based diagnosis and treatment of obstructive sleep apnea. Chest. 2010 Aug;138(2):257-63. doi: 10.1378/chest.09-0577. Epub 2010 Feb 19. PMID 20173052
- [Background] Rosen CL, Auckley D, Benca R, Foldvary-Schaefer N, Iber C, Kapur V, Rueschman M, Zee P, Redline S. A multisite randomized trial of portable sleep studies and positive airway pressure autotitration versus laboratory-based polysomnography for the diagnosis and treatment of obstructive sleep apnea: the HomePAP study. Sleep. 2012 Jun 1;35(6):757-67. doi: 10.5665/sleep.1870. PMID 22654195
- [Background] Mitchell RB, Pereira KD, Friedman NR. Sleep-disordered breathing in children: survey of current practice. Laryngoscope. 2006 Jun;116(6):956-8. doi: 10.1097/01.MLG.0000216413.22408.FD. PMID 16735907
- [Background] Roland PS, Rosenfeld RM, Brooks LJ, Friedman NR, Jones J, Kim TW, Kuhar S, Mitchell RB, Seidman MD, Sheldon SH, Jones S, Robertson P; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: Polysomnography for sleep-disordered breathing prior to tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jul;145(1 Suppl):S1-15. doi: 10.1177/0194599811409837. Epub 2011 Jun 15. PMID 21676944
- [Background] Kirk V, Baughn J, D'Andrea L, Friedman N, Galion A, Garetz S, Hassan F, Wrede J, Harrod CG, Malhotra RK. American Academy of Sleep Medicine Position Paper for the Use of a Home Sleep Apnea Test for the Diagnosis of OSA in Children. J Clin Sleep Med. 2017 Oct 15;13(10):1199-1203. doi: 10.5664/jcsm.6772. PMID 28877820
- [Background] Cho S, Ensari I, Weng C, Kahn MG, Natarajan K. Factors Affecting the Quality of Person-Generated Wearable Device Data and Associated Challenges: Rapid Systematic Review. JMIR Mhealth Uhealth. 2021 Mar 19;9(3):e20738. doi: 10.2196/20738. PMID 33739294
- [Background] Kannampallil T, Ma J. Digital Translucence: Adapting Telemedicine Delivery Post-COVID-19. Telemed J E Health. 2020 Sep;26(9):1120-1122. doi: 10.1089/tmj.2020.0158. Epub 2020 May 18. PMID 32427529
- [Background] Berry RB, Quan SF, Abreu AR. The AASM Manual for the Scoring of Sleep and Associated Events: Rules, Terminology, and Technical Specifications. 2.6 ed. Darien, IL: American Academy of Sleep Medicine; 2020.
- [Derived] Roman Rosado YD, Somayaji M, Stefanovski D, Uwah EA, Ward M, Tapia IE, Galion A, DelRosso LM, Davidson Ward SL, Cielo CM. Randomised trial of home sleep apnoea testing compared to in-lab polysomnography for the evaluation of obstructive sleep apnoea in children: rationale and study protocol. BMJ Open. 2025 Jun 24;15(6):e103315. doi: 10.1136/bmjopen-2025-103315. PMID 40555446